CLINICAL TRIAL: NCT05406219
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BAY 2395840 in Participants With Moderate Renal Impairment and in Healthy Male and Female Participants With Normal Renal Function
Brief Title: A Study to Learn How the Study Treatment BAY2395840 Moves Into, Through and Out of the Body, How Safe it is, and How it Affects the Body in Participants With Moderate Reduced Kidney Function and in Healthy Male and Female Participants With Normal Kidney Function
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuation of program.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 22044
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Neuropathic Pain; Renal Impairment; Healthy Volunteers
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: moderately impaired renal function (Experimental): Participants with moderately impaired renal function will receive a single dose of BAY2395840.
  Interventions: Drug: BAY2395840
- Group 2: normal renal function matched to Group 1 (Experimental): Participants with normal renal function matched to Group 1 will receive a single dose of BAY2395840.
  Interventions: Drug: BAY2395840
- Group 3: normal renal function aiming to balance out Group 2 (Experimental): Participants with normal renal function aiming to balance out Group 2 for the age and gender investigations will receive a single dose of BAY2395840.
  Interventions: Drug: BAY2395840

INTERVENTIONS:
Drug: BAY2395840 — Immediate release (IR) tablet, oral administration

SUMMARY:
Researchers are looking for a better way to treat people who have inflammatory conditions.

Inflammatory conditions may result from an increased activation of the body's natural defenses (the immune system) and are characterized by swelling, redness, heat, and pain.

The study treatment BAY2395840 is under development for use in inflammatory conditions. It works by blocking a protein, the B1 receptor, whose activation is involved in inflammatory responses.

The main purpose of this study is to learn how a single dose of BAY2395840 moves into, through and out of the body in participants with a moderate reduction of kidney function compared to matched participants with normal kidney function.

To answer this, the researchers will compare:

* the (average) total level of BAY2395840 in the blood (also known as AUC), and
* the (average) highest level of BAY2395840 in the blood (also known as Cmax) between the two groups of participants. The participants do not benefit from this study. However, the study will provide information on how to use BAY2395840 in later studies in people with inflammatory conditions. As some people with these conditions may also have kidney problems, this study is done in participants with moderate reduction of kidney function to characterize the use of BAY2395840 in this patient group.

All participants will take a single dose of BAY2395840 as tablets. Each participant will be in the study for up to 5 weeks. They will stay in-house for 4 days, including one treatment day. In addition, one visit before and one visit after the in-house phase to the study site is planned.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older, at the time of signing the informed consent.
* Participants who are - apart from renal function - overtly healthy for their age as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants with moderate renal impairment with an eGFR of 30 to 59 mL/min/1.73 m^2 (inclusive) according to the Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)
* Normal renal function, as assessed by estimated glomerular filtration rate (eGFR) based on serum creatinine at screening according to the modified Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI) formula: eGFR ≥90 mL/min/1.73 m^2. For participants with an age of 65 years and older, an eGFR of ≥ 60 mL/min/1.73 m^2 is acceptable.
* Body mass index (BMI) within the range 18 - 32 kg/m^2 (inclusive).
* Male and female participants had to use safe contraception, as defined by guidelines for contraception in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Medical disorder, condition or history of such that would impair the participant's ability to take part in or complete this study.
* Acute renal failure or acute nephritis within the past 2 years.
* Existing chronic diseases requiring medication (applicable only for Group 2 and Group 3 for those younger than 65 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-08-17 (Estimated); Study Completion 2023-10-12 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity (AUC) after single dose of BAY 2395840 | From pre-dose up to 72 hours post administration
  AUC(0-tlast) will be used as the main parameter if AUC cannot be reliably determined
Maximum observed drug concentration in measured matrix (Cmax) after single dose of BAY 2395840 | From pre-dose up to 72 hours post administration
Unbound area under the concentration vs. time curve from zero to infinity (AUCu) after single (first) dose of BAY 2395840 | From pre-dose up to 72 hours post administration
  AUC(0-tlast)u will be used as the main parameter if AUC cannot be reliably determined
Unbound maximum observed drug concentration in measured matrix (Cmax,u) after single dose of BAY 2395840 | From pre-dose up to 72 hours post administration

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From application of study intervention until follow-up Day 9

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.